CLINICAL TRIAL: NCT06054438
Title: Examining the Immunomodulatory and Health Improving Function of a Chinese Medicine Nutritional Supplement Cs4 on Immunity-related Disorders in the Post-COVID Era
Brief Title: Examining the Function of Cs4 on Post-COVID-19 Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor FENG Yibin, Professor, Director, The University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UW23-011; Innovation and Technology Fund (Other Grant/Funding Number: PRP/069/22FX)
Record Dates: First submitted 2023-09-25; First posted 2023-09-26 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A- having treatment at first stage (Other): 110 long-COVID patients will be divided into 2 groups (55 individuals per group).
  ⚫ Group A: 55 long-COVID patients (NO. 1- NO.55) Group B: 55 long-COVID patients (NO. 56- NO.110)
  Group distribution and treatment in a two-stage waitlist design: ⚫ First-stage clinical trial for 12 weeks:
  Group A (patients NO.1-55 will have treatment) Group B (patients NO.56-110 will have no Cs4 treatment on the waiting list)
  ⚫ Second-stage clinical trial for 12 weeks (After finishing the first-stage study): Group A (patients NO.1-55 will have no Cs4 treatment) Group B (patients NO.56-110 will have Cs4 treatment)
  Interventions: Other: Chinese medicine nutritional supplement Cs4
- Group B- having treatment at secondstage (Other): 110 long-COVID patients will be divided into 2 groups (55 individuals per group).
  ⚫ Group A: 55 long-COVID patients (NO. 1- NO.55) Group B: 55 long-COVID patients (NO. 56- NO.110)
  Group distribution and treatment in a two-stage waitlist design: ⚫ First-stage clinical trial for 12 weeks:
  Group A (patients NO.1-55 will have treatment) Group B (patients NO.56-110 will have no Cs4 treatment on the waiting list)
  ⚫ Second-stage clinical trial for 12 weeks (After finishing the first-stage study): Group A (patients NO.1-55 will have no Cs4 treatment) Group B (patients NO.56-110 will have Cs4 treatment)
  Interventions: Other: Chinese medicine nutritional supplement Cs4

INTERVENTIONS:
Other: Chinese medicine nutritional supplement Cs4 — Cs4 will be provided by Chinese Pharm, produced by GMP standard manufacturing. The intervention will be given according to the product instruction. Each capsule is 0.4g. According to the product sheet, adults should take 3-4 capsules daily as a way to nourish and strengthen the lungs and kidneys. In our study, the participants are people with long-COVID symptoms. Therefore, in order to achieve maximum efficacy, we will follow the directions and let participants take the maximum amount allowed by the product which is 4 capsules daily. Participants will take one capsule (each 400mg) 4 times a day, for a total of 1.6g. Treatment will last 12 weeks.

SUMMARY:
Cordyceps is a medicinal Chinese medicine. The benefits of cordyceps-related therapeutic action have been studied due to its anti-inflammation and immunomodulation features. Thus, Cordyceps may have efficacy against health problems in the post-COVID era. the Cs4 is a Chinese medicine nutritional supplement fermented by Cordyceps. This Project conducts a two-stage waitlist-controlled trial to examine the therapeutic effect of the Cs4 on long-COVID patients. 110 Patients will be recruited and divided into two groups. Each group contains 55 patients. In the first-stage clinical trial for 12 weeks, group A will have treatment while group B will have no Cs4 treatment. In the second-stage clinical trial for 12 weeks, group A will have no Cs4 treatment while group B will have Cs4 treatment. A 12-week follow-up will be conducted after the intervention of Cs4 for group A. The primary outcome will be the change from 0 to 12 weeks in symptom severity measured by self-declared modified COVID-19 Yorkshire Rehabilitation Scale (C19-YRSm). In our study, we intend to analyse the efficacy of Cs4 on the improvement of long Covid symptoms by using a comprehensive measurement to cover most symptoms, and be condition-specific. The secondary outcomes will include the change from 0 to 12 weeks of Insomnia Severity Index (ISI), Brief Fatigue Inventory Form, St. George's Respiratory Questionnaire (SGRQ), Hospital Anxiety and Depression Scale (HADS), and the Short Form 12 (SF12). Blood tests will be assessed for safety study. primary outcomes and secondary outcomes will be assessed at baseline (week 0) and week 12. The anticipated outcome of the study is to provide evidence of Cs4 in the improvement of long COVID symptoms. This project can serve to the development of a nutritional supplement for the management of post-COVID-related health problems.

DETAILED DESCRIPTION:
Research Methodologies Participants Setting This is a waitlist-controlled trial to examine the therapeutic effect of Cs4 on long-COVID patients, which are divided into two groups. The study will be conducted in the Specialist Clinical Centre for Teaching and Research (Sassoon Road), School of Chinese Medicine, The University of Hong Kong (HKU).

Inclusion Criteria

1. Male or female patients with age from 18 to 75 years old, who have been previously diagnosed with COVID-19 and recovered;
2. The self-declared post-COVID-19 Functional Status scale should be at least over 1;
3. The post-COVID symptoms have lasted at least 28 days after diagnosis;
4. Currently not taking any other orally administered Chinese medicine;
5. Negative COVID-19 antigen or nucleic acid test within 3 days prior to signing the consent form;
6. Voluntary participation in this clinical study. Exclusion Criteria

1. Inability to read and/or write Chinese or English; 2. Inability to communicate (e.g. with cognitive impairment) 3. Allergy to Cordyceps sinensis; 4. Pregnant or lactating women; 5. Impaired hepatic or renal function. Methods Participants will be recruited through the webpage of the School of Chinese Medicine, HKU. Clinical history and comprehensive examination will be performed during the first interview by registered Chinese Medicine practitioners or registered nurses who will be informed about the aims, procedure and nature of the study, and possible side effects of Cs4 and written consent will be obtained from each subject who agrees to get into the study. The participant will be also informed that they have the freedom to withdraw at any time during the study.

Study design This will be a waitlist-controlled trial in which participants will alternately receive the intervention of Cs4 for 12 weeks, followed by a 12-week follow-up. 110 long-COVID patients will be randomly divided into two groups (Group A and Group B). Randomisation will be carried out according to the computer- based Excel random number generator. An integer number between 1 and 110 will be assigned to each individual at random. Group A consists of individuals assigned integer numbers between 1 and 55. Group B consists of individuals assigned integer numbers between 56 and 110.

Intervention Cs4 will be provided by Chinese Pharm, produced by GMP standard manufacturing. The intervention will be given according to the product instruction. Each capsule is 0.4g. According to the product sheet, adults should take 3-4 capsules daily as a way to nourish and strengthen the lungs and kidneys. In our study, the participants are people with long-COVID symptoms. Therefore, in order to achieve maximum efficacy, we will follow the directions and let participants take the maximum amount allowed by the product which is 4 capsules daily. Participants will take one capsule (each 400mg) 4 times a day, for a total of 1.6g. Treatment will last 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with age from 18 to 75 years old, who have been previously diagnosed with COVID-19 and recovered;
2. The self-declared post-COVID-19 Functional Status scale should be at least over 1;
3. The post-COVID symptoms have lasted at least 28 days after diagnosis;
4. Currently not taking any other orally administered Chinese medicine;
5. Negative COVID-19 antigen or nucleic acid test within 3 days prior to signing the consent form;
6. Voluntary participation in this clinical study.

Exclusion Criteria:

1. Inability to read and/or write Chinese or English;
2. Inability to communicate (e.g. with cognitive impairment) 3. Allergy to Cordyceps sinensis;

4. Pregnant or lactating women; 5. Impaired hepatic or renal function.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
the change in symptom severity from 0 to 12 weeks measured by the modified COVID-19 Yorkshire Rehabilitation Scale (C19-YRSm) | will be assessed at baseline and 12 weeks.
  Symptom severity is one of the sub-scale of C19-YRSm. Range 0-78, with higher scores indicating greater impact of symptoms. C19-YRSm is the first validated scale describing post-COVID-19 symptoms and grading the severity of symptoms and functional disability.

SECONDARY OUTCOMES:
the change in Insomnia Severity Index (ISI) from 0 to 12 weeks | will be assessed at baseline and 12 weeks.
  To evaluate insomnia. Maximum values: 28, minimum values:0. Higher scores mean a worse outcome.
the change in Brief Fatigue Inventory Form (BFI) from 0 to 12 weeks | will be assessed at baseline and 12 weeks.
  To evaluate fatigue. Maximum values: 10, minimum values:0. Higher scores mean a worse outcome.
the change in St. George's Respiratory Questionnaire (SGRQ) from 0 to 12 weeks | will be assessed at baseline and 12 weeks.
  To evaluate respiratory symptoms. Maximum values: 100, minimum values:0. Higher scores mean a worse outcome.
the change in Hospital Anxiety and Depression Scale (HADS) from 0 to 12 weeks | will be assessed at baseline and 12 weeks.
  To evaluate anxiety and depression. Maximum values: 21, minimum values:0. Higher scores mean a worse outcome.
the change in Short Form 12 (SF12) from 0 to 12 weeks | will be assessed at baseline and 12 weeks.
  To evaluate overall quality of life. Maximum values: 100, minimum values:0. Higher scores mean better physical and mental health functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Yibin Feng, Doctor, Principal Investigator — The University of Hong Kong
Locations (1):
- The School of Chinese Medicine, HKU, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whitworth J. COVID-19: a fast evolving pandemic. Trans R Soc Trop Med Hyg. 2020 Apr 8;114(4):241-248. doi: 10.1093/trstmh/traa025. No abstract available. PMID 32198918
- [Background] Garg M, Maralakunte M, Garg S, Dhooria S, Sehgal I, Bhalla AS, Vijayvergiya R, Grover S, Bhatia V, Jagia P, Bhalla A, Suri V, Goyal M, Agarwal R, Puri GD, Sandhu MS. The Conundrum of 'Long-COVID-19': A Narrative Review. Int J Gen Med. 2021 Jun 14;14:2491-2506. doi: 10.2147/IJGM.S316708. eCollection 2021. PMID 34163217
- [Background] Chen J, Chan WM, Leung HY, Leong PK, Yan CTM, Ko KM. Anti-Inflammatory Effects of a Cordyceps sinensis Mycelium Culture Extract (Cs-4) on Rodent Models of Allergic Rhinitis and Asthma. Molecules. 2020 Sep 4;25(18):4051. doi: 10.3390/molecules25184051. PMID 32899766
- [Background] Han F, Dou M, Wang Y, Xu C, Li Y, Ding X, Xue W, Zheng J, Tian P, Ding C. Cordycepin protects renal ischemia/reperfusion injury through regulating inflammation, apoptosis, and oxidative stress. Acta Biochim Biophys Sin (Shanghai). 2020 Feb 3;52(2):125-132. doi: 10.1093/abbs/gmz145. PMID 31951250
- [Background] Klok FA, Boon GJAM, Barco S, Endres M, Geelhoed JJM, Knauss S, Rezek SA, Spruit MA, Vehreschild J, Siegerink B. The Post-COVID-19 Functional Status scale: a tool to measure functional status over time after COVID-19. Eur Respir J. 2020 Jul 2;56(1):2001494. doi: 10.1183/13993003.01494-2020. Print 2020 Jul. PMID 32398306
- [Background] Sivan M, Preston N, Parkin A, Makower S, Gee J, Ross D, Tarrant R, Davison J, Halpin S, O'Connor RJ, Horton M. The modified COVID-19 Yorkshire Rehabilitation Scale (C19-YRSm) patient-reported outcome measure for Long Covid or Post-COVID-19 syndrome. J Med Virol. 2022 Sep;94(9):4253-4264. doi: 10.1002/jmv.27878. Epub 2022 Jun 1. PMID 35603810